CLINICAL TRIAL: NCT04143932
Title: Multiple Myeloma Patient Registry - Prospective National Multi Center Prospective Study
Brief Title: Multiple Myeloma Turkish Prospective Patient Registry
Acronym: THD-MM-Reg
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Turkish Hematology Association (Other)
Responsible Party: Sponsor
Other Study IDs: THD-MM-Reg
Record Dates: First submitted 2019-10-27; First posted 2019-10-30 (Actual); Last update posted 2023-07-18 (Actual); Status verified 2023-07

CONDITIONS: Multiple Myeloma; Relapse Multiple Myeloma
Keywords: multiple myeloma; MM; Registry; Turkey
MeSH Terms: conditions — Multiple Myeloma

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 3 Years
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
This is a non-interventional, national, multi center, prospective multiple myeloma registry in Turkey

DETAILED DESCRIPTION:
In this study, approximately from 40 centers 1000 patients will be recruited. All patients will be followed-up till the study end.

All the laboratory results, treatment protocols and responses will be recorded and assessed with EORTC Multiple Myeloma Specific Quality of Life Multiple Myeloma Specific (MY-20) and EORTC Quality of Life-C30 questionnaires.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosed as multiple myeloma
* Patients signed informed consent form
* Patients received no more then 2 lines of therapy

Exclusion Criteria:

* Patients below 18 years old

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All patients diagnosed as multiple myeloma received maximum 2 lines of therapy will be included to this prospective registry.
Sampling Method: Probability Sample
Enrollment: 1000 (Estimated)
Dates: Start 2020-10-10 (Actual); Primary Completion 2024-12 (Estimated); Study Completion 2024-12 (Estimated)

PRIMARY OUTCOMES:
Overall Survival | [Time Frame: 5 Years]
  Time from the diagnosis to the death
Progression Free Survival | [Time Frame: 5 Years]
  Time from the initiation of treatment to the death from any cause or progression

CONTACTS AND LOCATIONS:
Overall Officials: Omur Gokmen Sevindik, Assoc. Prof., Principal Investigator — Medipol University Hospital
Locations (1):
- Medipol University, Istanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No